CLINICAL TRIAL: NCT04467320
Title: Addressing Elevated PTSD Symptoms in Young People in Care: A Randomised Feasibility Trial Across Social-care and Mental Health Services.
Brief Title: Recovery Learning for Adolescents After Traumatic Experiences
Acronym: RELATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of East Anglia (Other); King's College London (Other); University of Edinburgh (Other); University of Bristol (Other); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government)
Responsible Party: Principal Investigator, Sarah Halligan, Professor of Child and Family Mental Health, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274914
Record Dates: First submitted 2020-06-23; First posted 2020-07-13 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Post Traumatic Stress Disorder; PTSD; Trauma; Foster care; RCT; group
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either the online intervention group (Teaching Recovery Techniques) or the care-as-usual group. Any young people entering into the trial who live in the same household will be randomised together. If randomised to the TRT condition, each child will be offered participation in the next age-appropriate group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Receiving the Teaching Recovery Techniques intervention (delivered online).
  Interventions: Behavioral: Teaching Recovery Techniques
- Care-As-Usual Group (Active Comparator): Receiving care-as-usual.
  Interventions: Behavioral: Care as usual

INTERVENTIONS:
Behavioral: Teaching Recovery Techniques — Teaching Recovery Techniques is a 7-session group programme, with 5-sessions for the young person and 2-sessions for the carer. All sessions will be held online. The carer sessions are focused on psychoeducation around trauma and PTSD, as well as skills for supporting a young person through the intervention and with PTSD symptoms more broadly. The young person sessions are primarily focused on skill building and include: psychoeducation and understanding intrusive memories; intrusive images, worries and dreams; arousal, emotions, relaxation and coping; avoidance and triggers; and, memories.
  Arms: Intervention Group
Behavioral: Care as usual — In the care as usual arm, social workers will follow their standard care protocol for young people experiencing psychological distress. A typical response may include a referral to either the specialist local CAMHS or general CAMHS.
  Arms: Care-As-Usual Group

SUMMARY:
Most children who have been removed from their family home and placed under the care of a Local Authority have been exposed to many frightening experiences, including witnessing violence, not being fed or cared for, or being abused. These experiences can lead to significant emotional difficulties. One such difficulty is posttraumatic stress disorder (PTSD), which can involve symptoms like having constant "flashbacks" of scary experiences, and a constant feeling of being in danger. This can have a big effect on children's lives. Yet, it is still not clear how to help young people in care who are experiencing high PTSD symptoms.

One idea the researchers have is to use a group-based online programme which has successfully helped other young people who have been exposed to different kinds of stressful experiences (for example, war). To test whether this programme could help children in care too, the researchers first need to see whether social workers have the time to check in with a child about PTSD symptoms; whether young people and their carers are willing to be involved in a research project which will test out the treatment programme; and whether mental health workers might face any problems when delivering the programme. This project aims to answer these questions.

The researchers will train social workers to complete an 8-question interview with 10-17 year olds in care, which will measure symptoms of PTSD. If the young person is experiencing high symptoms, they will be invited to take part in a research project. If they would like to join the project, children will be randomly selected to take part in the online group programme, or be given care-as-usual. The group programme involves the young person taking part in five weekly meetings held online, where they will learn skills to reduce their distress, and be supported to work through their difficult memories. Their carers will also take part in two online meetings which will teach them how to support their young person.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing elevated PTSS (using a standard cut-off score of =/> 17 on the 8-item Child Revised Impact of Events Scale; CRIES-8).
* Living in any care residence (with the exception of those living with a biological parent).
* Access to appropriate technology to engage in the online sessions and can do so in a quiet and private space.

Exclusion Criteria:

* A diagnosis of psychosis.
* Current and active serious suicidal ideations.
* A moderate to severe learning disability.
* Currently receiving direct therapeutic mental health support.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Child and Adolescent Trauma Screen (CATS) | 6 months
  Self-report DSM-5 post-traumatic stress disorder (PTSD) symptom measure. Scores range from 0-60, with greater scores indicating greater symptom severity.

SECONDARY OUTCOMES:
Child Revised Impact of Events Scale (CRIES-8) | 6 months
  Self-report post-traumatic stress disorder (PTSD) symptom screening tool. Symptom scores range from 0-40, with higher scores indicating greater symptom severity.
Child PTSD Symptom Scale (CPSS-5) Interview Schedule | 6 months
  DSM-5 PTSD diagnostic interview. Symptoms range from 0-80, with higher scores indicating greater symptom severity.
Inventory of Parent and Peer Attachment (IPPA) | 6 months
  Self-report measure of young person's perception of their relationship with their carer. Scores range from 28-140, with lower scores indicating greater relationship difficulties.
Strengths and Difficulties Questionnaire (SDQ) | 6 months
  Self-report and carer-report measure of internalising and externalising difficulties. There are 5 subscales each with scores ranging from 0-10. The total difficulties score is calculated by summing 4 of the sub-scales to give a score between 0-40. The greater the total score, the greater the difficulties experienced.
Short Mood and Feelings Questionnaire (SMFQ) | 6 months
  Self-report and carer-report depression questionnaire. Scores range from 0-26, with higher scores indicating more depressive symptoms.
Child Health Utility 9D (CHU9D) | 6 months
  Self-report measure of health-related quality of life. Scores range from 9-45, with higher scores indicating greater difficulties.
Parent Trauma Response Questionnaire - support style subscale (PTRQ) | 6 months
  Carer-report measure of their support style. Scores range from 0-30, with higher scores indicating greater difficulties.
Child and Adolescent Trauma Screen (carer report) | 6 months
  Carer-report young person PTSD symptom scale. Symptom scores range from 0-60, with higher scores indicating greater symptom severity.

OTHER OUTCOMES:
Focus groups and 1:1 semi-structured interviews | 2 months
  Qualitative measures carried out with young people, carers and service providers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hiller RM, Davis RS, Devaney J, Halligan SL, Meiser-Stedman R, Smith P, Stallard P, Kandiyali R, MacNeill S. Protocol for the RELATE trial: a feasibility and pilot randomised controlled trial of a low-intensity group intervention for young people in care with elevated posttraumatic stress symptoms. Pilot Feasibility Stud. 2021 Nov 13;7(1):204. doi: 10.1186/s40814-021-00936-7. PMID 34774093